CLINICAL TRIAL: NCT05644535
Title: Correlation Between Blood Biochemical Indicators and Cerebrospinal Fluid Gravity in Aged Patients
Brief Title: Cerebrospinal Fluid Gravity Correlation Analysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First People's Hospital of Chenzhou (Other)
Responsible Party: Principal Investigator, zhiming zhang, MD, Ph.D, First People's Hospital of Chenzhou
Other Study IDs: 202201
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Specific Gravity; Cerebrospinal Fluid
Keywords: Cerebrospinal fluid; Correlation Analysis; Lighter Specific Gravity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid of the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: Patients were aged 60-69 years
  Interventions: Diagnostic Test: Cerebrospinal fluid densitometry; Diagnostic Test: blood routine examination; Diagnostic Test: Blood electrolyte examination
- Group B: Patients were aged 70-79 years
  Interventions: Diagnostic Test: Cerebrospinal fluid densitometry; Diagnostic Test: blood routine examination; Diagnostic Test: Blood electrolyte examination
- Group C: Patients were aged 80-89 years
  Interventions: Diagnostic Test: Cerebrospinal fluid densitometry; Diagnostic Test: blood routine examination; Diagnostic Test: Blood electrolyte examination
- Group D: Patient age > 90 years
  Interventions: Diagnostic Test: Cerebrospinal fluid densitometry; Diagnostic Test: blood routine examination; Diagnostic Test: Blood electrolyte examination

INTERVENTIONS:
Diagnostic Test: Cerebrospinal fluid densitometry — After obtaining the patient's cerebrospinal fluid specimen, the actual mass of the cerebrospinal fluid was measured by pipetting 1000 μL of cerebrospinal fluid specimen on an analytical balance using a pipette gun, and all specimens were measured three times and the average of the three times was taken as the final mass of 1000 μL of that specimen. After the mass measurement, the residual cerebrospinal fluid was disposed of as medical waste. The density of each specimen was obtained according to the density to mass conversion formula ρ=m/v.
Diagnostic Test: blood routine examination — After obtaining the patient's blood specimens, they were sent to the laboratory for blood routine examination.
Diagnostic Test: Blood electrolyte examination — After obtaining the patient's blood specimens, they were sent to the laboratory for blood electrolyte examination.

SUMMARY:
The purpose of this study was to measure cerebrospinal fluid density in aged patients and to see if there was a correlation between these factors and cerebrospinal fluid density by using the electronic medical record system to understand the patient's gender, blood glucose, blood biochemical electrolytes and blood levels.

DETAILED DESCRIPTION:
Hip joint injury is one of the common injuries in the elderly, and hip arthroplasty is a treatment method that allows patients to get out of bed and return to social life as soon as possible. Currently, the common position for hip arthroplasty is the lateral position; and combined spinal and epidural anesthesia or subarachnoid anesthesia is also the common anesthesia method for hip arthroplasty. In the lateral position, the patient's affected limb is often on top and the healthy limb is on the bottom; the healthy side position is also the usual position for hip arthroplasty. In this position, it may be optimal to use a lighter specific gravity local anesthetic drug because it tends to anesthetize only the upper affected limb and does not require a return to the supine position after anesthesia due to changes in the plane of block, minimizing pain and hemodynamic fluctuations during anesthesia and position changes.

Currently, light specific gravity is more of a concept. Because in the available data, only the range of cerebrospinal fluid density of ordinary healthy adults is available, there is little literature and data to describe and analyze what the cerebrospinal fluid density of elderly patients actually is. Therefore, when we administer subarachnoid anesthesia to elderly patients, we cannot determine whether the dispensed local anesthetic drug is a light specific gravity.

In this study, we intend to collect cerebrospinal fluid from elderly patients who underwent hip arthroplasty under combined lumbar and rigid anesthesia or subarachnoid anesthesia, and measure the cerebrospinal fluid density in elderly patients, and observe whether there is a correlation between the above factors and cerebrospinal fluid density through the electronic medical record system to understand the patient's gender, blood glucose, blood biochemical electrolytes and routine blood levels; thus, we can better guide the use of lighter specific gravity drugs in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Receiving combined spinal and epidural anesthesia or subarachnoid anesthesia ASA Ⅰ or Ⅱ patients No significant neurological pathology No recent history of cerebral infarction No recent history of cerebral hemorrhage No central nervous system inflammation No spinal inflammatory disease No history of spinal surgery Patients who have given pre-operative informed written consent

Exclusion Criteria:

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Selected aged patients who had hip arthroplasty in our hospital between December 2022 and May 2023
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Cerebrospinal fluid density | baseline (before anesthesia)
  After obtaining the mass of cerebrospinal fluid, the density was calculated from ρ=m/v

SECONDARY OUTCOMES:
Blood sugar | baseline (before anesthesia)
  Plasma glucose level
Plasma K+ concentration | baseline (before anesthesia)
  Plasma K+ concentration
Plasma Cl- concentration | baseline (before anesthesia)
  Plasma Cl- concentration
WBC | baseline (before anesthesia)
  Leukocyte concentration in blood
Neutrophil concentration in blood | baseline (before anesthesia)
  Neutrophil concentration in blood
Lymphocyte concentration in blood | baseline (before anesthesia)
  Lymphocyte concentration in blood
C-reactive protein (CRP) | baseline (before anesthesia)
  C-reactive protein concentration in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Zhiming Zhang, Chenzhou, Hunan, China